CLINICAL TRIAL: NCT04514822
Title: Quantitative Evaluation of Metastatic Lymph Nodes With Dynamic 2-[18F]Fluoro-2-deoxy-glucose (18F-FDG) Positron Emission Tomography/Computed Tomography in Patients With Esophageal Squamous Cell Carcinoma
Brief Title: Quantitative Evaluation of Metastatic Lymph Nodes With Dynamic 18F-FDG PET/CT in Patients With ESCC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fifth Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ZDWY.FZYX.006
Record Dates: First submitted 2020-05-10; First posted 2020-08-17 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2020-02

CONDITIONS: Esophageal Squamous Cell Carcinoma; Positron Emission Tomography
Keywords: Esophageal squamous cell carcinoma; metastatic lymph nodes; positron emission tomography; glucose metabolic rate
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- N0 stage (Other): patients without malignant lymph nodes
  Interventions: Diagnostic Test: Dynamic PET
- Non-N0 stage (Other): patients with malignant lymph nodes
  Interventions: Diagnostic Test: Dynamic PET

INTERVENTIONS:
Diagnostic Test: Dynamic PET — After transmission CT scan for subsequent PET data attenuation correction, continual dynamic clinical PET scans were performed in a single bed position immediately after 18F-FDG intravenously injection (210 ± 30 MBq) in list mode for 60 minutes in supine position, dynamic 48 time frames PET/CT imaging was obtained.And then underwent whole body static PET scan.
  Other Names: Static PET

SUMMARY:
Currently, static scans are commonly used for Positron Emission Tomography/Computed Tomography (PET/CT) examination in the literature. Accordingly, functional images of 2-[18F]fluoro-2-deoxy-glucose (18F-FDG) Positron Emission Tomography/Computed Tomography (PET/CT) with dynamic scans can be more sensitive to detect metastatic lymph node, since the introduction of temporal dynamic variables would provide more imaging quantification than conventional static scans. The purpose of this study is to provide the dynamic 18F-FDG PET/CT imaging for esophageal squamous cell carcinoma (ESCC) patient to quantify the difference between malignant lymph nodes (MLN) and benign lymph nodes (BLN).

DETAILED DESCRIPTION:
Esophageal cancer is one of the most aggressive malignancies in the world, which accounted for an estimated 572,034 new cases and 508,585 deaths in 2018 worldwide. The incidence and mortality of esophageal cancer is ranked first in China and esophageal squamous cell carcinoma (ESCC) is the main histological subtype of esophageal cancers in China. Correct preoperative evaluation of whether the tumor has reached any lymph nodes is important for management. Various methods have been used to detect primary and lymph node metastases in esophageal cancer patients, including computed tomography (CT), endoscopic examinations, and endoscopic ultrasonography (EUS). However, even such advanced imaging modalities do not always reliably identify lymph node metastasis prior to surgical resection and pathological examination.

The appearance of lymph nodes with morphological imaging procedures is classified by their shape, size, density and, if applied, contrast enhancement. BLN usually tend to have a fatty hilum, an oval shape and frequently do not measure more than 1 cm in the short axis diameter. However, the use of size as the most important criterion for differentiation of benign and malignant lymph nodes has limitations: small metastases without an increase in lymph node size are frequently missed. Positron emission tomography (PET)/computed tomography (CT) is increasingly used as single "one stop shop" method, which the combination of morphological and functional imaging represents the optimal approach for lymph node staging and general staging. A radioactive tracer，2-[18F]fluoro-2-deoxy-glucose (18F-FDG) currently used is based on the increased glucose metabolism, which may be reported with semiquantitative standard uptake value (SUV). Routinely, 18F-FDG is intravenous injected and PET/CT scan is performed after 60 min. The static imaging in differentiation of inflammatory from MLN may be problematic. Because inflammatory lymph nodes goes along with an increase in glucose metabolism, and thus may manifest increased 18F-FDG uptake. It was reported that PET-CT sensitivity and specificity for the detection of loco-regional metastases were moderate, but sensitivity and specificity were reasonable for distant metastases. Many researchers found there is a correlation between the 18F-FDG uptake and time. In malignancy, the uptake of FDG uptake continues to increase for several hours after FDG injection whereas such prolonged period of FDG uptake is rare in inflammatory/infectious or normal tissues. Shum et al ever assessed clinical usefulness of dual-time FDG PET/CT in esophageal squamous cell carcinoma, which turned out the sensitivity of FDG PET-CT in detecting the primary ESCC with combination of early maximum standard uptake value (SUVmax) ≥2.5 or retention index (RI) ≥10% was 96.2%. However, for loco-regional lymph node detection, there was no significant difference using dual-time 18F-FDG PET/CT assessment. Dynamic 18F-FDG PET/CT allows quantitative assessment of lesion in vivo by using a Patlak model to obtain the influx constant (Ki), and the glucose metabolic rate (MRglu). The purpose of the study is to determine whether the dynamic 18F-FDG PET/CT imaging (0-60 min) add additional value in differentiation MLN from BLN.

ELIGIBILITY:
Inclusion Criteria:

·Patients who were pathologically confirmed ESCC at Sun Yet-sen Fifth Affiliated Hospital.

Exclusion Criteria:

* diabetes mellitus
* fasted glucose level ≥ 11.0 mmol/L
* breast feeding
* pregnancy and clustrophobia.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Ki comparison between MLNs and BLNs | 60 minutes
  Ki of each MLN and BLN were calculated and compared
MRglu comparison between MLNs and BLNs | 60 minutes
  MRglu of each MLN and BLN were calculated and compared
SUVmax comparison between MLNs and BLNs | 60 minutes
  SUVmax of each MLN and BLN were calculated and compared
SUVmax 60/30 comparison between MLNs and BLNs | 60 minutes
  SUVmax 60/30 of each MLN and BLN were calculated and compared

SECONDARY OUTCOMES:
Ki comparison from PTs between N0 and non-N0 stage | 60 minutes
  Ki of each primary tumor between N0 and non-N0 stagewere calculated and compared
MRglu comparison from PTs between N0 and non-N0 stage | 60 minutes
  MRglu of each primary tumor between N0 and non-N0 stagewere calculated and comparedtumor were calculated.
SUVmax comparison from PTs between N0 and non-N0 stage | 60 minutes
  SUVmax of each primary tumor between N0 and non-N0 stagewere calculated and comparedtumor were calculated.
SUVmax 60/30 comparison from PTs between N0 and non-N0 stage | 60 minutes
  SUVmax 60/30 of each primary tumor between N0 and non-N0 stagewere calculated and compared

OTHER OUTCOMES:
Sensitivity | 60 minutes
  The sensitivity for each parameter in differentiating malignant and benign lymph nodes were evaluated
Specificity | 60 minutes
  The specificity for each parameter in differentiating malignant and benign lymph nodes were evaluated
Accuracy | 60 minutes
  The accuracy for each parameter in differentiating malignant and benign lymph nodes were evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Hong Shan, Ph.D, Study Chair — Fifth Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The Fifth Affiliated Hospital, Sun Yat-sen University, Zhuhai, Guangdong, China

IPD SHARING:
Plan to Share IPD: No